CLINICAL TRIAL: NCT02889185
Title: Multimodal Imaging in Central Serous Chorioretinopathy
Acronym: IMO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P/2015/249
Record Dates: First submitted 2016-08-31; First posted 2016-09-05 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Central Serous Chorioretinopathy
Keywords: Optical Coherence Tomography; Retinal camera
MeSH Terms: conditions — Central Serous Chorioretinopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adaptative optics retinal camera (Experimental)
  Interventions: Device: RTX1 IMAGIN EYE retinal camera

INTERVENTIONS:
Device: RTX1 IMAGIN EYE retinal camera — In addition to the routine examination including OCT, an imaging using RTX1 IMAGIN EYE retinal camera will be performed.

SUMMARY:
This study aims to assess the contribution of the multimodal imaging, combining a routine examination using Optical Coherence Tomography (OCT) with an imaging procedure using adaptive optics retinal camera.

This is a feasibility study with a limited number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form
* Beneficiary/affiliated to French social security/social healthcare
* Active ou chronic Central Serous Chorioretinopathy on at least one eye
* Absence of other known ophthalmological pathology or of any ophthalmological conditions revealed during the examination

Exclusion Criteria:

* Legal incapacity or limited legal capacity
* Predictable poor adherence
* Subject without health insurance
* Pregnant or breatfeeding women
* Sujet étant dans la période d'exclusion d'une autre étude ou prévue par le "fichier national des volontaires"
* Presence of transparent medium opacity damaging images quality
* Previous photosensitivity
* Recent treatment with PhotoDynamic Therapy (PDT)
* Use of drugs inducing photosensitivity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-04; Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
Workability of images of RTX1 IMAGIN EYE retinal camera | day 1
  Two readings of the images captured with adaptative optics retinal camera and assessment of their workability in routine care.

CONTACTS AND LOCATIONS:
Overall Officials: Maher Saleh, MD PhD, Principal Investigator — CHU Besançon
Locations (1):
- CHU Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No